CLINICAL TRIAL: NCT04601402
Title: A Phase I/Ib Study to Evaluate the Safety, Tolerability, Biological and Clinical Activities of GEN-001 in Combination With Avelumab in Patients With Advanced Solid Tumors Who Have Progressed During or After Treatment With Anti-PD-(L)1 Therapy
Brief Title: GEN-001 (Live Biotherapeutic Product) and Avelumab Combination Study for Patients With Solid Tumors Who Have Progressed on Anti-PD-(L)1 Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genome & Company (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: [GNC] GEN001-101
Record Dates: First submitted 2020-10-13; First posted 2020-10-23 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Dose Escalation: Seqeuntial Group Assignment, Dose Expansion: Parallel Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN-001 with avelumab (Experimental): Dose Escalation Cohort includes patients with advanced or metastatic solid tumors who have progressed on at least two lines of approved therapy for their histological subtypes which includes an anti-PD-1 or anti-PD-L1 based therapy (as mono or combination) will be enrolled. 3 or 6 patients will be enrolled per escalating or de-escalating dose levels.
  Dose Expansion Cohort includes patients with advanced or metastatic NSCLC, SCCHN, and UC who have progressed on at least two lines of approved therapy for their histological subtypes which includes an anti-PD-1 or anti-PD-L1 based therapy (as mono or combination)will be enrolled.
  Interventions: Drug: GEN-001; Drug: Avelumab

INTERVENTIONS:
Drug: GEN-001 — The capsules taken by mouth once a daily. Each capsule will contain ≥ 1x10^11 colony-forming units (CFU)
Drug: Avelumab — 800 mg given by intravenous (IV) infusion once every 2 weeks
  Other Names: Bavencio

SUMMARY:
This is a phase I/Ib, first-in-human (FIH), open-label, dose escalation and dose expansion study to evaluate the safety and tolerability, biological and clinical activities of GEN-001 in patients with locally advanced or metastatic solid tumors who have progressed on at least two lines of approved therapy for their histological subtypes which includes an anti-PD-1 or anti-PD-L1 based therapy (as mono or combination), when administered as combined with avelumab.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have adequate organ functions as defined in the protocol
* Negative childbearing potential
* Have ability to swallow and retain oral medication and no clinically significant gastrointestinal abnormalities
* Patients with diseases for which no curative therapies are available, and who have progressed on at least two lines of approved therapy for their histological subtypes which includes an anti-PD-1 or anti-PD-L1 based therapy (as mono or combination)
* Disease progression on anti-PD-(L)1 based therapy (as monotherapy or combination therapy) and must meet criteria for acquired resistance as defined in the protocol
* Patients who have completely recovered from any clinically significant AEs that occurred during prior immunotherapy
* Estimated life expectancy of at least 3 months
* Objective evidence of disease progression at baseline (Dose Escalation)
* Histologically or cytologically confirmed, unresectable, locally advanced, or metastatic NSCLC, SCCHN, and UC (Dose Expansion)
* Measurable disease as per RECIST v1.1 defined as at least 1 lesion (Dose Expansion)

Exclusion Criteria:

* Have experienced primary resistance to anti-PD-(L)1 based therapy
* Has experienced a toxicity that led to permanent discontinuation of prior anti-PD-(L)1 based therapy or other immunotherapies
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Current use of immunosuppressive medication at time of study entry
* Have an active infection requiring antibiotics, antifungal or antiviral agents or have received a course of antibiotics within the previous 4 weeks of starting study treatment
* Has received a live vaccine within 4 weeks of starting of study treatment
* Known history of, or any evidence of active, non-infectious pneumonitis
* Prior solid organ or allogeneic stem cell transplantation
* Has had any investigational or anti-tumor treatment within 4 weeks or 5 half-life periods of starting study treatment, had any major surgeries within 4 weeks of starting study treatment
* Has received proton pump inhibitors (PPIs) within 2 weeks prior to dosing study treatments
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has clinically significant (i.e., active) cardiovascular disease
* Has known history of uncontrolled intercurrent illness
* Has any psychiatric condition that would prohibit the understanding or rendering of informed consent or that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of Adverse Events | 1 years
  Assessed as per CTCAE v5.0
Dose Escalation: Incidence of Laboratory abnormalities | 1 years
  Assessed as per CTCAE v5.0
Dose Escalation: Incidence of dose-limiting toxicity (DLT) | 1 Cycle (one cycle = 28 days)
  To evaluate the safety and tolerability of GEN-001 in combination with avelumab
Dose Expansion: To assess objective response (OR) of GEN-001 in patients with advanced or metastatic solid tumors, when administered as combined with avelumab. | 2 years
  Confirmed OR per RECIST v1.1 by the Investigator

SECONDARY OUTCOMES:
Objective Response (OR) | 1 years
  Assessed according to RECIST v1.1
Duration of response (DoR) | up to 2 years
  Assessed according to RECIST v1.1
Progression-free survival (PFS) | up to 2 years
  Assessed according to RECIST v1.1
Overall Survival (OS) | up to 2 years
Incidence of Adverse Events | up to 2 years
  Assessed as per CTCAE v5.0
Incidence of Laboratory Abnormalities | up to 2 years
  Assessed as per CTCAE v5.0
irOR (Immune-related Objective Response) | up to 2 years
  Assessed according to irRECIST

OTHER OUTCOMES:
Ctrough | up to 2 years
  Ctrough for PK parameter
ADA | up to 2 years
  Anti-Drug Antibodies(ADA) for Immunogenicity
Microbiota | up to 2 years
  fecal samples will be collected for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No